CLINICAL TRIAL: NCT06594315
Title: Assessing Brain Metabolism Using 1H MRS With Deuterated Glucose
Brief Title: Assessing Brain Metabolism Using MRS With Deuterated Glucose
Status: Active, not recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 22922; NCI-2022-08563 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Glioma
Keywords: Glucose Metabolism
MeSH Terms: conditions — Glioma | interventions — Glucose; Magnetic Resonance Spectroscopy; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort 1: Healthy Controls: Twenty healthy controls for will have 2H-glucose metabolism in measured for development of robust strategy in optimizing acquisition parameters.
  Interventions: Drug: Deuterated Glucose; Procedure: Magnetic Resonance Imaging (MRI); Procedure: Blood Sample; Procedure: MR spectroscopy (MRS)
- Cohort 2: Glioma participants (Single Time point): Thirty participants with glioma who may or may not have received prior treatment for testing the optimized imaging protocol developed in Cohort 1.
  Interventions: Drug: Deuterated Glucose; Procedure: Magnetic Resonance Imaging (MRI); Procedure: Blood Sample; Procedure: MR spectroscopy (MRS)
- Cohort 3: Glioma participants (Multiple Time points): Thirty participants who will receive non-investigational treatment for glioma enrolled to test the evaluation for treatment induced metabolic changes at baseline and post- non-investigational treatment.
  Interventions: Drug: Deuterated Glucose; Procedure: Magnetic Resonance Imaging (MRI); Procedure: Blood Sample; Procedure: MR spectroscopy (MRS)

INTERVENTIONS:
Drug: Deuterated Glucose — Given orally
  Other Names: Hydrogen gas (H2) glucose; [6,6'-2H2] glucose
Procedure: Magnetic Resonance Imaging (MRI) — Imaging procedure performed at University of California, San Francisco
  Other Names: MRI
Procedure: Blood Sample — Capillary blood from the fingertip
Procedure: MR spectroscopy (MRS) — Imaging procedure performed at University of California, San Francisco
  Other Names: MRS

SUMMARY:
This study will investigate the use of Hydrogen 1 (1H) magnetic resonance spectroscopy (MRS) with deuterated glucose (2H-glucose) to detect dynamic glucose uptake in the brain.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

1. To define the most appropriate imaging parameters of 1H MRS for obtaining deuterium-labeled glucose metabolism (Cohorts 1 and 2).
2. To evaluate treatment induced metabolic changes after the administration of 2H-glucose in participants with glioma (Cohort 3).

OUTLINE:

Participants with and without glioma will be evaluated to develop a robust strategy for obtaining 2H-glucose metabolism in twenty healthy participants (cohort 1) and thirty participants with glioma (cohort 2), while the remaining thirty glioma participants will be studied at baseline and after completion of non-investigational therapy (cohort 3).

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be >= 18 years old

   * Cohort 1: Healthy controls
   * Cohort 2: Participants with histological proven glioma who have evidence of evaluable disease (with contrast enhancing lesion or non-enhancing lesion > 4 cc) based on a prior MR scan, Karnofsky performance status of >=70 and life expectancy > 4 weeks.
   * Cohort 3: Participants with histologically proven glioma who will be undergoing any treatment, Karnofsky performance status of >=70 and life expectancy > 12 weeks.
2. Participants must not have any significant medical illness that in the investigator's opinion cannot be adequately controlled with appropriate therapy, would compromise the subject's ability to participate in this study or any disease that will obscure toxicity or dangerously impact response to the imaging agent.
3. Participants must not have a history of any other cancer unless they are in complete remission and have been off all therapy for that disease for a minimum of 3 years.
4. Participants must not be pregnant or breast-feeding. Persons of childbearing potential are required to obtain a negative serum or urine pregnancy test within 14 days of the scan. Effective contraception (men and women) must be used in subjects of childbearing potentials.
5. Participants must sign an informed consent indicating that they are aware of the investigational nature of the study

Exclusion Criteria:

Participants must be excluded from participating in this study if they are not able to comply with the study and/or follow-up procedures.

1. Participants exceeding the weight limitations of the scanner (300 pounds)
2. Inability to lie still for the entire imaging time (e.g., cough, severe arthritis, etc.)
3. Inability to complete the study due to other reasons (severe claustrophobia, MR incompatible medical implants or devices, inability to comply with pre-procedure fasting, etc.)
4. Pre-examination blood glucose level of > 120 mg/dL as measured by point of care finger stick blood glucose test prior to MR examination.
5. Participants, either healthy volunteers (recruited for cohort 1) or participants with glioma (for cohorts 2 &3), have history of diabetes mellitus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults and adult patient referrals from the UCSF Neuro-Oncology Service and Department of Neurological Surgery.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-07-20 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Signal-to-noise ratio (Cohort 1 & 2) | Day of imaging (1 day)
  The signal-to-noise ratio (SNR) in metabolite concentrations will be calculated and compared on a voxel-by-voxel basis and via summary parameters (mean, median, and max) from the regions of interest (ROIs) of the anatomic and metabolic lesions on the imaging scan. Peaks with SNR > 5.0 are considered detectable
Mean difference in metabolite concentrations (Cohort 1 & 2) | Day of imaging (1 day)
  Mean difference in metabolite concentrations of 2H labeling of these metabolites will be calculated and compared on a voxel-by-voxel basis and via summary parameters (mean, median, and max) from the ROIs of the anatomic and metabolic lesions.
Mean difference in fractional enrichment (Cohort 1 & 2) | Day of imaging (1 day)
  Mean difference in fractional enrichment of 2H labeling of these metabolites will be calculated and compared on a voxel-by-voxel basis and via summary parameters (mean, median, and max) from the ROIs of the anatomic and metabolic lesions.
Mean metabolic turnover over time (Cohort 3) | Up to 21 days after the completion of non-investigational treatment
  Estimates of the extent of change over time following non-investigational treatment obtained at the baseline and one repeated after receiving treatment will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Li, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No